CLINICAL TRIAL: NCT01806870
Title: Immune Enhancement for Immunological Non-responders to ART
Acronym: IMMUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David M. Guidot, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00062730; 1R34HL117351-01 (NIH)
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: HIV
Keywords: HIV; ART
MeSH Terms: interventions — Zinc; S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional Supplements Zinc and SAMe (Experimental): Each subject will receive 1600mg of SAMe per day Men subjects will receive 30mg Zinc Women subjects will receive 25mg Zinc
  Interventions: Dietary Supplement: Zinc and SAMe

INTERVENTIONS:
Dietary Supplement: Zinc and SAMe — If a subject has side effects their dose of Zinc will be reduced. SAMe will remain the same dose.

SUMMARY:
The purpose of this study is to see if taking two nutritional supplements, zinc and SAMe (S-adenosylmethionine), can improve lung health and immune function in persons with HIV. You are being asked to volunteer because you have HIV (Human Immunodeficiency Virus) and you take anti-retroviral therapy (ART) medications.

DETAILED DESCRIPTION:
There will be up to eleven study visits and three telephone visits. All study procedures are for research purposes. All study subjects will receive the nutritional supplements zinc and SAMe.

During the study you will be asked to answer questions about your alcohol use and smoking history. You will have exhaled breath tests, blood draws, physical exams, and bronchoscopies. Your medical records will be reviewed during the study. If you are a woman of childbearing age, a urine pregnancy test will be done at each study visit.

Visit 1 (screening visit): This visit will last about 2 hours. At this visit you will:

* Have a physical exam
* Review your medical history
* Review your medications
* Have blood drawn
* Have a urine pregnancy test for women of child-bearing age
* Complete a survey about your alcohol use and smoking history.
* Discuss and schedule a bronchoscopy for the next visit You may not be eligible to continue in the study if the blood work done at visit one is not within normal limits or if you are pregnant. A study team member will contact you to let you know if you do or do not qualify to participate in the remainder of the study.

Visit 2: This visit will last about 6 hours and will take place at the Hospital. At this visit you will:

* Have a physical exam
* Have blood drawn
* Have a urine pregnancy test for women of child-bearing age
* Do an exhaled breath test
* Have a bronchoscopy
* Receive nutritional supplements and education

Treatment: The nutritional supplements zinc and SAMe will be given to you by the study team at visit 2. You will be asked to take the tablets once a day.

If you experience upset stomach, abdominal cramps, diarrhea, or other uncomfortable side effects, we will reduce the amount of the nutritional supplements. If you are unable to tolerate the nutritional supplements, you will be withdrawn from the research study.

Visits 3, 4, and 5 -Telephone Contact: You will receive a telephone call at one, two, and three weeks after visit 2 to ask you how you are tolerating the study supplements. If you are experiencing side effects such as upset stomach, abdominal cramps, or diarrhea, we will instruct you to decrease the dose of the supplements.

Visits 6, 7, and 8 (months one, two, and three): These visits will last about 30 minutes and will be scheduled two months apart. At this visit you will:

* Have blood drawn
* Have a urine pregnancy test for women of child-bearing age
* Do an exhaled breath test
* Answer questions about how you are tolerating the nutritional supplements
* Receive nutritional supplements and education

If your exhaled breath test is at goal at visit 6, you will continue to take the dietary supplements for one year from this point forward. If your exhaled breath test is not at goal at visit 6, you will be asked to return for visit 7. If your exhaled breath test is at goal at visit 7, you will continue to take the dietary supplements for one year from this point forward. If your exhaled breath test is not at goal at visit 7, you will be asked to return for visit 8. You will be asked to take the nutritional supplements for one year from this point forward.

Visits 9 through 13: These visits will last about 30 minutes and will be scheduled two months apart.

At this visit you will:

* Have blood drawn
* Have a urine pregnancy test for women of child-bearing age
* Answer questions about how you are tolerating the nutritional supplements
* Receive nutritional supplements and education

Visit 14: This is the final study visit. It will last about 6 hours and will take place at the Hospital. At this visit you will:

* Have a physical exam
* Have blood drawn
* Have a urine pregnancy test for women of child-bearing age
* Do an exhaled breath test
* Have a bronchoscopy procedure
* Return unused nutritional supplements

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects living with HIV-1 infection who have been on anti-retroviral therapy (ART) for a minimum of 18 months and:

  * are followed longitudinally for their HIV healthcare in one of the study sites in Atlanta or Seattle
  * meet criteria for immunological non-responsiveness as defined by adherence to ART and cluster of differentiation 4 (CD4) count <350 despite adequate retroviral suppression.
* 2. Ability to give informed consent.

Exclusion Criteria:

1. Documented history of cirrhosis or a total bilirubin ≥ 2.0 mg/dL.
2. Documentation of left ventricular ejection fraction < 40% or myocardial infarction within the past 6 months.
3. End-stage renal disease requiring dialysis or a serum creatinine ≥ 2 mg/dL.
4. Spirometry with Forced vital capacity (FVC) or Forced expiratory volume in 1 second (FEV1) < 70% of predicted value.
5. Diabetes
6. Known or possible pregnancy or attempting to become pregnant.
7. BMI < 17
8. Age < 21
9. Parkinson's disease: these are all b/c the SAMe risks sections states that these pts will not qualify
10. Bipolar disorder
11. Bleeding disorders such as thrombocytopenia or significant gastrointestinal bleeding within the past year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Immune Enhancement for Immunological Non-responders to ART | First 6 months
  Optimize the dosing of dietary zinc and SAMe that restores redox balance and zinc bioavailability in the airways of a cohort of HIV-infected individuals who are 'immunological non-responders'

CONTACTS AND LOCATIONS:
Overall Officials: David Guidot, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Hospital- Ponce De Leon Clinic, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2013-02-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT01806870/ICF_000.pdf